CLINICAL TRIAL: NCT05350449
Title: Loving Kindness Meditation Among Adults 50 Years and Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Nirmala Lekhak, PhD, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNLV-2022-148
Record Dates: First submitted 2022-04-08; First posted 2022-04-28 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Loneliness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loving kindness meditation (Experimental): Loving-kindness meditation is a contemplative practice that focuses on developing compassion for oneself and others through mindfulness. Participants will be shown the recorded loving-kindness training video during the first week of the intervention. Participants will be encouraged to use the mp3 device with guided meditation recording to practice mindfulness meditation for 20-25 minutes every day for 30 days. We will also provide participants with a diary to record their daily meditation experiences. There will be weekly check in. At 60 days we will do a follow-up data collection.
  Interventions: Behavioral: Loving-kindness Meditation
- Waitlist control (No Intervention): The arm will eventually get the intervention.

INTERVENTIONS:
Behavioral: Loving-kindness Meditation — Loving-kindness meditation is a type of mindfulness practice where the focus is on love/compassion and kindness for self and others. The guided meditation will be provided via recording device. The intervention is 4 week long.
  Other Names: mindfulness practice
  Arms: Loving kindness meditation

SUMMARY:
The goal of this clinical trial is to test the feasibility and acceptability of loving-kindness meditation among adults 50 years and older. It will also examine the benefits of this intervention and compare the outcomes between two groups (intervention and wait-list control).

DETAILED DESCRIPTION:
The main aim of the research is to assess the feasibility and acceptability of the Loving-kindness meditation intervention among adults 50 years or older. It will also examine the intervention's preliminary impact on loneliness, self-compassion, cognitive function, and psychological well-being. The study will use a randomized controlled trial with waitlist control.

ELIGIBILITY:
Inclusion Criteria:

• Adults 50 years or older living in Southern Nevada

Exclusion Criteria:

• Cognitive or language barrier that would make it difficult to understand and sign the informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirmala Lekhak, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Loving Kindness Meditation: Loving-kindness meditation is a contemplative practice that focuses on developing compassion for oneself and others through mindfulness. Participants will be shown the recorded loving-kindness training video during the first week of the intervention. Participants will be encouraged to use the mp3 device with guided meditation recording to practice mindfulness meditation for 20-25 minutes every day for 30 days. We will also provide participants with a diary to record their daily meditation experiences. There will be weekly check in. At 60 days we will do a follow-up data collection.
  Loving-kindness Meditation: Loving-kindness meditation is a type of mindfulness practice where the focus is on love/compassion and kindness for self and others. The guided meditation will be provided via recording device. The intervention is 4 week long.
  22 participants
- Waitlist Control: The arm will eventually get the intervention.
  23 participants
Period: Overall Study
Arm/Group | Loving Kindness Meditation | Waitlist Control
Started | 28 | 31 (We had to move 2 participants to control group because after randominzation they said that time might work better for control group.)
Completed | 24 | 23
Not Completed | 4 | 8
Not completed — Withdrawal by Subject | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loving Kindness Meditation | Waitlist Control | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.1 (6.2) | 71.5 (6.9) | 72.8 (6.6)
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.1 (6.2) | 71.5 (6.9) | 72.8 (6.6)
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.1 (6.2) | 71.5 (6.9) | 72.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 2 | 6
  White | 20 | 25 | 45
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 28 | 31 | 54
Loneliness [Mean (Standard Deviation); unit: units on a scale] | 4.6 (1.6) | 4.7 (1.9) | 4.7 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Loneliness
Description: A 3-item modified UCLA loneliness scale will be used to measure loneliness. The scores on this scale range from 3 to 9, the highest scores indicative of a higher level of loneliness. We will measure loneliness at baseline, post-intervention and 2 follow-up periods to measure the change in loneliness level because of the loving-kindness meditation intervention.
Time Frame: baseline, immediately post-intervention, and week 4 and week 8 post intervention (follow-up periods).
Population: Baseline population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loving Kindness Meditation | Waitlist Control
Number analyzed (Participants) | 28 | 31
units on a scale
  Baseline | 4.64 (1.64) | 4.65 (1.85)
  Post-Intervention: number analyzed (Participants) | 28 | 26
  Post-Intervention | 4.82 (1.68) | 4.62 (1.69)
  Week 4 follow up: number analyzed (Participants) | 27 | 20
  Week 4 follow up | 4.56 (1.48) | 4.55 (1.82)
  Week 8 follow up: number analyzed (Participants) | 27 | 22
  Week 8 follow up | 4.74 (1.85) | 4.09 (1.63)

2. Primary Outcome: Change in Self-compassion
Description: A 12-item Self-compassion Short form Scale by Kirsten Neff will be used to measure self-compassion. The scores on this scale rages from 1-5. The highest scores are indicative of better self-compassion. We will measure self-compassion at baseline and post-intervention periods to measure the change in self-compassion because of the loving-kindness meditation intervention.
Time Frame: baseline, immediately post-intervention, and week 4 and week 8 post intervention.
Population: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Loving Kindness Meditation | Waitlist Control
Number analyzed (Participants) | 28 | 31
units on a scale
  Baseline | 3.5 (0.63) | 3.62 (0.87)
  Post-intervention: number analyzed (Participants) | 28 | 26
  Post-intervention | 3.29 (0.75) | 3.61 (0.92)
  Week 4 follow-up: number analyzed (Participants) | 26 | 20
  Week 4 follow-up | 3.43 (0.66) | 3.82 (0.98)
  Week 8 follow-up: number analyzed (Participants) | 26 | 20
  Week 8 follow-up | 3.6 (0.75) | 4.03 (1.02)

3. Secondary Outcome: Change in Anxiety
Description: A 4-item PROMIS Emotional Distress: Anxiety Scale will be used to measure anxiety. The scores on this scale range from 4 to 20, the highest scores indicative of a higher feeling of anxiety. We will measure anxiety at baseline and post-intervention periods to measure the change in anxiety level because of the loving-kindness meditation intervention.
Time Frame: baseline, immediately post-intervention, and week 4 and week 8 post intervention.
Population: Some of participants did not enter the data for some timelines.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loving Kindness Meditation | Waitlist Control
Number analyzed (Participants) | 28 | 31
units on a scale
  baseline: number analyzed (Participants) | 27 | 28
  baseline | 8.33 (3.34) | 8.61 (3.87)
  post intervention: number analyzed (Participants) | 28 | 26
  post intervention | 8.89 (3.2) | 9.54 (3.85)
  week 4 follow-up: number analyzed (Participants) | 25 | 21
  week 4 follow-up | 7.76 (3.26) | 8.33 (3.95)
  week 8 follow-up: number analyzed (Participants) | 26 | 22
  week 8 follow-up | 8.54 (4.01) | 7.5 (3.64)

4. Secondary Outcome: Change in Depressive Symptoms
Description: A 10-item Center for Epidemiologic Studies Short Depression Scale will be used to measure depressive symptoms. The scores on this scale range from 10 to 40, the highest scores indicative of a higher feeling of depression. We will measure depressive symptoms at baseline and post-intervention periods to measure the change in depressive symptoms because of the loving-kindness meditation intervention.
Time Frame: baseline, immediately post-intervention, and week 4 and week 8 post intervention.
Population: not all participants entered data for each timeline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loving Kindness Meditation | Waitlist Control
Number analyzed (Participants) | 28 | 31
units on a scale
  baseline: number analyzed (Participants) | 25 | 28
  baseline | 16.72 (5.32) | 17.04 (5.65)
  post-intervention: number analyzed (Participants) | 28 | 26
  post-intervention | 18.21 (4.79) | 18.12 (6.34)
  week 4 follow-up: number analyzed (Participants) | 27 | 21
  week 4 follow-up | 16.74 (5.01) | 16.14 (6.11)
  week 8 follow-up: number analyzed (Participants) | 27 | 22
  week 8 follow-up | 18.07 (7.09) | 15.50 (5.73)

ADVERSE EVENTS:
Time Frame: Adverse events and deaths were **not monitored**, (e.g., "All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed").
Description: Adverse events and deaths were **not monitored**. So no participants were at risk.
Arm/Group | Loving Kindness Meditation | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT05350449/Prot_SAP_ICF_000.pdf